CLINICAL TRIAL: NCT06360562
Title: Reconnecting to Ourselves and Others in Virtual Meetings (ROOM)- Resilience Training in Virtual Reality
Brief Title: Reconnecting to Ourselves and Others in Virtual Meetings (ROOM)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daphne Holt, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P002418
Record Dates: First submitted 2023-08-29; First posted 2024-04-11 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Mood Disorders; Anxiety Disorders; Psychotic Disorders
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Resilience Training (Experimental): A 6 1-hour session group based intervention to deliver mindfulness, metallization, and self-compassion.
  Interventions: Behavioral: Resilience Training

INTERVENTIONS:
Behavioral: Resilience Training — Behavioral group-based intervention delivering mindfulness, metallization, and self-compassion skills.

SUMMARY:
This study aimed to determine the feasibility and acceptability of delivering Resilience Training in multi-user virtual reality.

ELIGIBILITY:
Inclusion criteria for college student participants:

1. 18-30 years old
2. Enrolled in an undergraduate program

Inclusion criteria for healthcare provider participants:

1. At least 18 years old
2. Employed in the healthcare field with some direct patient contact

Exclusion Criteria:

1. Inability to provide informed consent
2. Not proficient in English
3. Acute symptoms of a psychiatric illness needing immediate care (such as acute psychotic symptoms, current suicidality, serious active alcohol or substance use, marked deterioration in functioning over the prior month) determined by self-report that necessitates close monitoring or inpatient or partial hospitalization.
4. Enrolled in current psychotherapy with frequency of more than once per month

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Discomfort with Others | Before the intervention, 6 weeks later, and 6 months later
  Discomfort with others is measured on a brief scale rated on a Likert scale of 1-5, asking three questions, how frequently someone feels discomfort with others, how intensely they feel it, and a multiple choice selection of reasons they may feel discomfort with others. Higher ratings indicate more discomfort with others.
Intervention Feasibility and Acceptability | Before the intervention, 6 weeks later, and 6 months later
  This measure includes participant attendance, with more attendance of the intervention indicating better feasibility and acceptability.
Penn Emotion Recognition Test | Before the intervention, 6 weeks later, and 6 months later
  The Penn Emotion Recognition Test (ER-40) is a 15-minute computer task which involves identifying the emotion (sadness, anger, etc.) expressed by a variety of face images with 5 possible options, was used to measure emotion recognition ability. The total score ranges from 0-40, with individual sub-scores for happy, sad, angry, fearful, and neutral expressions.
Stop Distance Paradigm | Before the intervention, 6 weeks later, and 6 months later
  The Stop Distance Paradigm is a reliable way to measure ones personal space. The larger the number, the larger the person stands from others. This scale is rated by centimeters from zero (no personal space) to as many as the person chooses. This task was done in person, through Zoom, and in virtual reality.

SECONDARY OUTCOMES:
Beck Depression Inventory | Before the intervention, 6 weeks later, and 6 months later
  The Beck Depression Inventory (BDI) is a 21-item self-report assessment obtaining ratings of one's level of depression on a Likert scale of 0-63, with higher scores indicating more depressive symptoms.
Spielberger State-Trait Anxiety Inventory | Before the intervention, 6 weeks later, and 6 months later
  The Spielberger State-Trait Anxiety Inventory (STAI) is a 20-item self-report scale obtaining ratings of one's anxiety, both those that are trait like and ongoing, and those that are state like and temporary. Scores range from 0-120, with higher scores indicate higher levels of anxiety symptoms.
Prodromal Questionnaire- Brief | Before the intervention, 6 weeks later, and 6 months later
  The Prodromal Questionnaire- Brief (PQ-B) is a 21-item self-report survey assessing psychotic experiences such as common delusional experiences (e.g. paranoia, grandiosity, ideas of reference) and perceptual aberrations (e.g. experiences of being controlled, mind reaching, etc.). and distress related to them. Each item is scored on a 0 to 5 scale. The total score is rated across the 21 items ranging between 0 and 105 with higher scores indicating more severe psychotic experiences.
Connor-Davidson Resilience Scale | Before the intervention, 6 weeks later, and 6 months later
  The Connor-Davidson Resilience Scale (CD-RISC) is a 25-item self-report scale obtaining ratings of one's level of coping and emotional resilience. It is rated on a scale of 0-100, with higher scores indicate one has more coping skills and more emotional resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared with investigator permission.

REFERENCES:
- [Derived] Holt DJ, DeTore NR, Aideyan B, Utter L, Vinke L, Johnson DS, Zimmerman J, Dokholyan KN, Burke A. Enhancing social functioning using multi-user, immersive virtual reality. Sci Rep. 2025 Jan 22;15(1):2790. doi: 10.1038/s41598-024-84954-4. PMID 39843493